CLINICAL TRIAL: NCT01861275
Title: Obstructive Sleep Apnea as a Risk Factor for Ischaemic Stroke , a Prospective Study
Brief Title: Ischaemic Stroke and Sleep Apnea in Northern Part of Finland
Status: Completed | Type: Observational
Sponsor: University of Oulu (Other)
Responsible Party: Sponsor
Other Study IDs: 36/2013; 36/2013 (Other: Oulu university hospital); 36/2013 UO (Other: Oulu university hospital)
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Sleep Apnoea; Cerebral Palsy
Keywords: osa; cerebral palsy; thrombolysis in cerebral palsy; sleep registration
MeSH Terms: conditions — Sleep Apnea Syndromes; Cerebral Palsy; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Nasal CPAP: We want to study the nasal-cpap treatment and it's compliance in sleep apnea patients with ischaemic stroke.
  Interventions: Device: Nasal CPAP
- no Nasal CPAP: No nasal-cpap in sleep apnea patients with ischaemic stroke.

INTERVENTIONS:
Device: Nasal CPAP — Nasal CPAP treatment for obstructive sleep apnoea
  Groups: Nasal CPAP

SUMMARY:
Obstructive sleep apnoea is a risk factor for ischaemic stroke. study hypothesis: In prospective study the investigators want to know how many ischaemic stroke patients have sleep apnoea and does thrombolysis play a role in severity of osa in six months follow up.

DETAILED DESCRIPTION:
In prospective study the investigators include all over 18 years old patients who came to emergency room for ischaemic stroke. Exclusion criteria is not able to co-operate or need for intensive care unit.The investigators shall take 100 control patients who have ischaemic stroke and no thrombolysis and 100 study patients who will have thrombolysis. The investigators do sleep registration during hospital staying within 2 days after patients have felt ill.Follow-up registration will be done after 6 months at home.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old patients that have cerebral palsy and are able to participate to the study.

Exclusion Criteria:

* no co-operation and need for intensive care unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: residents of Oulu university hospital area. consecutive patient sampling
Sampling Method: Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2013-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
cerebral palsy events and severity of osa | from six months to twenty four months
  in prospective study outcome measure is severity of osa in 6months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Tarja Saaresranta, Md PhD, Study Director — University hospital of Turku
Locations (1):
- Oulu university hospital,department of neurology, Oulu, Northern Finland, Finland

IPD SHARING:
Plan to Share IPD: Yes
Write a paper.

REFERENCES:
- [Derived] Huhtakangas JK, Saaresranta T, Vahanikkila H, Huhtakangas J. Nocturnal hypoxemia and central apneas increase mortality, but not recurrent ischemic events after ischemic stroke. Sleep Med. 2022 Sep;97:1-9. doi: 10.1016/j.sleep.2022.05.014. Epub 2022 May 23. PMID 35679775
- [Derived] Huhtakangas JK, Huhtakangas J, Bloigu R, Saaresranta T. Unattended sleep study in screening for sleep apnea in the acute phase of ischemic stroke. Sleep Med. 2020 Jan;65:121-126. doi: 10.1016/j.sleep.2019.08.002. Epub 2019 Aug 8. PMID 31751906
- [Derived] Huhtakangas JK, Saaresranta T, Bloigu R, Huhtakangas J. The Evolution of Sleep Apnea Six Months After Acute Ischemic Stroke and Thrombolysis. J Clin Sleep Med. 2018 Dec 15;14(12):2005-2011. doi: 10.5664/jcsm.7524. Erratum In: J Clin Sleep Med. 2020 May 15;16(5):837-838. doi: 10.5664/jcsm.8428. PMID 30518443
- [Derived] Huhtakangas JK, Huhtakangas J, Bloigu R, Saaresranta T. Prevalence of sleep apnea at the acute phase of ischemic stroke with or without thrombolysis. Sleep Med. 2017 Dec;40:40-46. doi: 10.1016/j.sleep.2017.08.018. Epub 2017 Oct 7. PMID 29221777